CLINICAL TRIAL: NCT04633993
Title: Effectiveness of Implementation of a Patient-centered Self-management Program in Patients With Hypertensive Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Cardinal Tien Hospital (Other)
Responsible Party: Principal Investigator, Mei-Chen Lee, RN, PhD, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTH-108-3-1-106
Record Dates: First submitted 2020-10-23; First posted 2020-11-18 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Hypertensive Nephropathy; Self-management; Self-efficacy; Mental Health Wellness 1
Keywords: hypertension; hypertensive nephropathy; chronic kidney disease; end-stage kidney disease,; patient-centered,; self-management program
MeSH Terms: conditions — Hypertensive Nephropathy; Hypertension; Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCSMP (Experimental): Patient-centered self-management program for patients with hypertensive nephropathy into 4 units, including: Unit 1: hypertensive nephropathy brief introduction and complications. Unit 2: dietary precautions for patients with hypertensive nephropathy. Unit 3: medication treatments for patients with hypertensive nephropathy. Unit 4: the content included stress management (emotional control, spiritual support). This program was implemented in small groups with 5-10 patients. This study used patient-centered self-management group activity manual as the tool. The group activities with 4 units lasting for 400 minutes were expected to be designed. The group activities were expected to last for 4 weeks and be implemented once per week and 100 minutes per time (including: 90 minutes of group discussion and 5-10 minutes of video-waring).
  Interventions: Behavioral: PCSMP
- Usual Care (No Intervention): Routine care.

INTERVENTIONS:
Behavioral: PCSMP — This study divided the patient-centered self-management manual for patients with hypertensive nephropathy into 4 units, including: Unit 1: hypertensive nephropathy brief introduction and complications. Unit 2: dietary precautions for patients with hypertensive nephropathy. Unit 3: medication treatments for patients with hypertensive nephropathy. Unit 4: the content included stress management (emotional control, spiritual support). This program was implemented in small groups with 5-10 patients. This study used patient-centered self-management group activity manual as the tool. The group activities with 4 units lasting for 400 minutes were expected to be designed. The group activities were expected to last for 4 weeks and be implemented once per week and 100 minutes per time (including: 90 minutes of group discussion and 5-10 minutes of video-waring).
  Other Names: Usual Care
  Arms: PCSMP

SUMMARY:
This study is a 2-years project. The year 1 project: to assess the effectiveness of implementation of the program in patients with HN. The experimental research design of 2×2 randomized controlled trial with pre and post-testing will be adopted. A total of 70 subjects will be enrolled, and 35 subjects will be randomized into the control group (conventional program) and experimental group (patient-centered self-management program), respectively, using the single-blind design. Firstly, this study will collect the pretest data of the control group and experimental group. The data to be collected include physiological indicators, physical and psychological health, self-efficacy, self-management, and satisfaction, etc. The experimental group will receive the 4-week intervention of program after the pre-test. This study will assess the effectiveness of intervention 1 month later. This study will use generalized estimating equation (GEE) to collect the longitudinal data and test the effectiveness of implementation of program in patients with HN at different time points (after 1, 3, and 6 months). It is expected that the completion of this research project may help improve the effective disease control in the care for patients with HN in Taiwan and improve self-management of disease. Hopefully, the incidence of patients with dialysis can be significantly reduced and the progression into ESRD in patients can be effectively delayed. Moreover, this study also intends propose specific suggestions about the care of patients with HN for industry, government, and academia.

DETAILED DESCRIPTION:
Since population aging is accompanied by chronic diseases. Hypertension is a type of chronic disease, and poor to control the symptoms of hypertension may accelerate the progression of renal function into hypertensive nephropathy (HN) and ultimately lead to dialysis. 2017 annual report on kidney disease in Taiwan published by The Taiwan Society of Nephrology showed that among the comorbidities experienced by new patients before the 1year dialysis, hypertension ranked the first (89.5%). In Taiwan, the prevalence and incidence of end-stage renal disease (ESRD) both are ranked high in the world, which has an impact on the aspects of individual, family, society, etc. and jeopardizes the financial situation of the government's national health insurance. Therefore, in order to effectively reduce the incidence of ESRD and delay the progression of HN, the implementation of a patient-centered self-management program may effectively reduce medical costs and improve patients' quality of life. This study is a 2-years project. The year 1 project to assess the effectiveness of implementation of the program in patients with HN. The experimental research design of 2×2 randomized controlled trial with pre and post-testing will be adopted. A total of 70 subjects will be enrolled, and 35 subjects will be randomized into the control group (conventional program) and experimental group (patient-centered self-management program), respectively, using the single-blind design. Firstly, this study will collect the pretest data of the control group and experimental group. The data to be collected include physiological indicators, physical and psychological health, self-efficacy, self-management, and satisfaction, etc. The experimental group will receive the 4-week intervention of program after the pre-test. This study will assess the effectiveness of intervention 1 month later. This study will use G power statistical analysis to calculate the sample size and use SPSS/Windows 20.0 for recording and statistical analysis. For the statistical analysis methods, this study will use repeated measure ANOVA to analyze the effectiveness of intervention. The year 2 project is to extend the year 1 research project. This study will use generalized estimating equation (GEE) to collect the longitudinal data and test the effectiveness of implementation of program in patients with HN at different time points (after 1, 3, and 6 months). It is expected that the completion of this research project may help improve the effective disease control in the care for patients with HN in Taiwan and improve self-management of disease. Hopefully, the incidence of patients with dialysis can be significantly reduced and the progression into ESRD in patients can be effectively delayed. Moreover, this study also intends propose specific suggestions about the care of patients with HN for industry, government, and academia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypertensive nephropathy and chronic kidney disease stage 3b to 5.
* Clear consciousness and could communicate in Chinese and Taiwanese
* Age 20 years old the above.

Exclusion Criteria:

* End-stage kidney disease who have undergone dialysis treatment (hemodialysis, peritoneal dialysis)
* Clinical diagnosis of diabetic nephropathy
* Diagnosed as mental illness (severe depression, schizophrenia) and cognitive dysfunction

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Hypertensive nephropathy self-management instrument (HN-SM) | 1st month, 3th month, and 6th month after recruited.
  The HN-SM: This scale is measured for evaluating the self-management of patients with hypertensive nephropathy in the past week. This scale is composed of 29 items in total, including 4 subscales: self-integration (10 questions), problem-solving (10 questions), seeking social support (5 questions), and compliance behavior (4 questions). This scale used four-point Likert scale for scoring: 1 point for "never", 2 point for "sometimes", 3 point for "often", and 4 point for "always". The total score ranged from 29 to 116 points. The reliability and validity of Cronbach'α was 0.77-0.92. The higher the total score, the better the patients with hypertensive nephropathy self-management.

SECONDARY OUTCOMES:
World Health Organization-5 Well Being Index (WHO-5) | 1st month, 3th month, and 6th month after recruited.
  WHO-5: This scale is measured for evaluating the physical and mental health status of patients with hypertensive nephropathy in the past week. This scale is a five-item questionnaire. This scale used six-point Likert scale for scoring: The scoring included 0 point for "at no time", 1 point for "sometimes", 2 point for "less than half time", 3 point for "more than half a time", 4 point for "most of the time", and 5 point for "all of the time". The total score ranges from 0 to 25 points. The Cronbach's α value of this scale is .87. Patients whose total score is lower than 13 points or whose answer to any of the 5 items is 0 to 1 point are recommended to receive the test of severe depression scale.
The hypertensive nephropathy self-efficacy instrument (HN-SE) | 1st month, 3th month, and 6th month after recruited.
  HN-SE: This study used this scale to test the level of self-confidence in disease self-management of patients with hypertensive nephropathy in the past week.This scale is a 25-item questionnaire. This scale used four-point Likert scale for scoring: The scoring included 0 point for "totally unsure" to 10 point for "very sure". The total score ranged from 0 to 250 points. The reliability and validity of Cronbach'α was 0.84-0.90. The higher the total score, the higher the level of self-confidence control of a disease self-management of patients with hypertensive nephropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Chen Lee, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Cardinal Tien Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Varleta P, Tagle R. A feared combination: Hypertension and chronic kidney disease. J Clin Hypertens (Greenwich). 2019 Jan;21(1):102-104. doi: 10.1111/jch.13432. Epub 2018 Nov 14. No abstract available. PMID 30427110
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Hypertension. 2018 Jun;71(6):1269-1324. doi: 10.1161/HYP.0000000000000066. Epub 2017 Nov 13. No abstract available. PMID 29133354
- [Background] Aryee C, Owiredu WK, Osei-Yeboah J, Owusu-Dabo E, Laing EF, Owusu IK. An Analysis of Anthropometric Indicators and Modifiable Lifestyle Parameters Associated with Hypertensive Nephropathy. Int J Hypertens. 2016;2016:6598921. doi: 10.1155/2016/6598921. Epub 2016 Sep 27. PMID 27774313
- [Background] Lin CC, Wu CC, Wu LM, Chen HM, Chang SC. Psychometric evaluation of a new instrument to measure disease self-management of the early stage chronic kidney disease patients. J Clin Nurs. 2013 Apr;22(7-8):1073-9. doi: 10.1111/j.1365-2702.2011.04048.x. Epub 2012 May 30. PMID 22642723
- [Background] Chow CK, Teo KK, Rangarajan S, Islam S, Gupta R, Avezum A, Bahonar A, Chifamba J, Dagenais G, Diaz R, Kazmi K, Lanas F, Wei L, Lopez-Jaramillo P, Fanghong L, Ismail NH, Puoane T, Rosengren A, Szuba A, Temizhan A, Wielgosz A, Yusuf R, Yusufali A, McKee M, Liu L, Mony P, Yusuf S; PURE (Prospective Urban Rural Epidemiology) Study investigators. Prevalence, awareness, treatment, and control of hypertension in rural and urban communities in high-, middle-, and low-income countries. JAMA. 2013 Sep 4;310(9):959-68. doi: 10.1001/jama.2013.184182. PMID 24002282
- [Background] Nguyen NT, Douglas C, Bonner A. Effectiveness of self-management programme in people with chronic kidney disease: A pragmatic randomized controlled trial. J Adv Nurs. 2019 Mar;75(3):652-664. doi: 10.1111/jan.13924. Epub 2019 Feb 14. PMID 30537153
- [Background] Wu SFV, Lee MC, Hsieh NC, Lu KC, Tseng HL, Lin LJ. Effectiveness of an innovative self-management intervention on the physiology, psychology, and management of patients with pre-end-stage renal disease in Taiwan: A randomized, controlled trial. Jpn J Nurs Sci. 2018 Oct;15(4):272-284. doi: 10.1111/jjns.12198. Epub 2017 Dec 20. PMID 29266792
- [Derived] Lee MC, Wu SV, Lu KC, Wang WH, Chen YY, Tai CY. Effect of Patient-Centered Self-Management Program on Blood Pressure, Renal Function Control, and the Quality of Life of Patients With Hypertensive Nephropathy: A Longitudinal Randomized Controlled Trial. Biol Res Nurs. 2022 Apr;24(2):216-225. doi: 10.1177/10998004211061877. Epub 2021 Dec 29. PMID 34964363
- [Derived] Lee MC, Wu SV, Lu KC, Wang WH, Chen YY, Chen HM. Effect of patient-centred self-management programme on mental health, self-efficacy and self-management of patients with hypertensive nephropathy: A randomised controlled trial. J Clin Nurs. 2021 Nov;30(21-22):3205-3217. doi: 10.1111/jocn.15825. Epub 2021 May 3. PMID 33942419